CLINICAL TRIAL: NCT02441192
Title: Cardiovascular and Cardiorespiratory Coupling After Different Types of Training and Detraining
Brief Title: Different Training (Aerobic, Resistance or Mixed) Physical Programs Affect to Physiological Responses (TRAINING2014)
Acronym: TRAINING2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Casimiro Javierre, Ph D, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: U.Barcelona
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Health Behavior
Keywords: physical training; aerobic training; resistance training
MeSH Terms: conditions — Health Behavior | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Training resistance (Experimental): After the baseline tests they were distributed in four randomized groups for the 6 weeks of training: aerobic (AT), resistance (RT), aerobic+resistance (AT+RT) and control (C).
  Interventions: Other: Training resistance
- Training aerobic (Experimental): After the baseline tests they were distributed in four randomized groups for the 6 weeks of training: aerobic (AT), resistance (RT), aerobic+resistance (AT+RT) and control (C).
  Interventions: Other: Training aerobic
- Training resistance+aerobic (Experimental): After the baseline tests they were distributed in four randomized groups for the 6 weeks of training: aerobic (AT), resistance (RT), aerobic+resistance (AT+RT) and control (C).
  Interventions: Other: Training resistance+aerobic

INTERVENTIONS:
Other: Training resistance — After the baseline tests they were distributed in four randomized groups for the 6 weeks of training: aerobic (AT), resistance (RT), aerobic+resistance (AT+RT) and control (C).
  Arms: Training resistance
Other: Training aerobic — After the baseline tests they were distributed in four randomized groups for the 6 weeks of training: aerobic (AT), resistance (RT), aerobic+resistance (AT+RT) and control (C).
  Arms: Training aerobic
Other: Training resistance+aerobic — After the baseline tests they were distributed in four randomized groups for the 6 weeks of training: aerobic (AT), resistance (RT), aerobic+resistance (AT+RT) and control (C).
  Arms: Training resistance+aerobic

SUMMARY:
Background. The cardiovascular and cardiorespiratory coupling (CVCRC), focusing to recognize the synergies of standard or modified physiology that promote healthy. The investigators aim to study the effects of different training modalities and detraining on CVCRC.

Methods. 32 young males were distributed in four randomized training groups: aerobic (AT), resistance (RT), aerobic plus resistance (AT+RT) and control (C). They were tested before, after the training (6 weeks) and after the detraining (3 weeks) through a graded maximal test. A principal component (PC) analysis of the time series of selected cardiovascular and cardiorespiratory variables was performed to evaluate the CVCRC. The PC1 coefficient of congruence in the 3 experimental conditions (before, after training and after detraining) was calculated for each group.

DETAILED DESCRIPTION:
The study of the cardiovascular and cardiorespiratory coupling (CVRC) is a hot topic in the medical literature focused to recognize the synergies that are present in healthy physiology [7, 8]. Several effects as aging [9], diseases [8] or mental state interventions [10] on cardiorespiratory coupling have been investigated, however, although its potential interest, there are no studies on the effects of training programs and detraining.

Two main types of training programs (aerobic- AT and resistance- RT) have been widely investigated by their important and different physiological effects [11]. Its combination (AT+RT), has been recently recommended with health purposes for extensive types of population [12-14].

The physiological effects of aerobic training programs has been traditionally evaluated through the cardiorespiratory reserve and the detection of maximal or threshold subsystem variables [1]. As a complex adaptive system (CAS), the human organism acts as an indivisible and integrated whole that cannot be reduced to the sum of its subsystems functions [2]. In this CAS the cardiovascular and cardiorespiratory subsystems are interdependent and interact in a dynamic and nonlinear way, i.e. non-proportional, which needs to be approached through nonlinear models [3], the study of time series and complex systems (CS) methodologies [4]. As the CAS enter every new situation with an existing set of capabilities [5] and exchange continuously information with their environment her/his behavior is unique and unexpected at short term (weeks, months) [6], the usual duration of common training programs.

In order to study the couplings and coordination between multiple variables in CAS, CS approaches propose the detection of the so-called order parameters, collective or coordinative variables, because they capture the order or coordination of the system [3, 15]. The principal component (PC) analysis is a common statistical technique that has been used to recognize such coordinative variables in a vast domain of biological research fields like: motor control [16], brain dynamics [17], DNA replication [18] or protein folding [19]. The PC analysis reduces the data dimension of highly coupled systems extracting the smallest number of components that account for most of the variation in the original multivariate data and summarize it with little loss of information. PCs are extracted in decreasing order of importance so that the first PC accounts for as much of the variation as possible and each successive component accounts for a little less [20]. The number of PCs reflects the dimensionality of the system, being a decrease of the number of PCs indicative of a major coupling (less dimensions) and vice-versa. The number of PCs changes when the system suffers a nonlinear change, i.e. a qualitative or coordinative reconfiguration. The PCs technique applied to kinematic variables has been successfully used to study the effects of motor learning processes [16], but has not been applied yet to study training effects on physiological variables.

The aim of this research was to investigate the dimensional changes of the CVCRC before and after a period of 6 weeks of different training modalities (AT, RT and AT+RT) and 3 weeks after detraining in healthy young men.

Material and Methods Participants. To determine the sample size a power analysis was performed. Using an effect size of d = .80, alfa < .05, power (1 - beta) = .95, with three repeated windows, we estimated a sample size = 32 [21]. Thirty-two healthy physically active males, physical education students (age 21.2 ± 2.4 y., height of 177.1 ± 0.66 cm, mean body mass 71.0 ± 5.1 kg and mean body -mass index 22.6 ± 1.7 kg·m-2) with no sport specialization but engaged in a wide range of aerobic activities at least three times a week volunteered to participate in this study. After the baseline tests they were distributed in four randomized groups for the 6 weeks of training: aerobic (AT), resistance (RT), aerobic+resistance (AT+RT) and control (C).

Procedure. Participants completed a standard medical questionnaire to confirm their healthy status and signed an informed consent form. All experimental procedures were approved by the local bio-ethics committee and were carried out in accordance with the ethical guidelines laid down in the Helsinki Declaration. After the baseline cardiorespiratory testing and maximal strength and power tests (see below) they followed 3 times a week their assigned specific training program:

1. AT group (n = 8): they pedalled 60 min at 60% of their individual maximum workload (60% Wmax). This workload was increased by 5% weekly unless the participant was unable to keep the pace throughout the session. Heart rate was monitored during all the sessions.
2. RT group (n = 8): they performed twice a 30 min strength circuit[14]. Forty per cent of 1RM for the upper body (i.e., squat, chest press, shoulder press, triceps extension, biceps curl, pull-down [upper back]), and 60% for the lower body (quadriceps extension, leg press, leg curls [hamstrings], and calf raise) were used as starting weights. They allowed the participants a maximum of 12 repetitions which included a slow controlled movement (2s up and 4s down). The resting period between exercises was 2 min. Workloads were adjusted weekly, with resistance being increased as needed (typically 5 up to 10%) if the participant was able to lift the weight comfortably (i.e., more than 12 repetitions).
3. AT+RT group (n = 8): they pedalled at 60% Wmax during 30 min and performed once the strength circuit (as R group).
4. C group (n = 8): continued with their usual activities, without any special training.

Cardiorespiratory testing. The incremental cycling test (Excalibur, Lode, Groningen, Netherlands) started at 0W and the workload increased 20W/min until exhaustion participants could not keep the prescribed cycling frequency of 70rpm during more than 5 consecutive seconds. All tests were performed in a well-ventilated lab; the room temperature was 23ºC and the relative humidity 48%, with variations of no more than 1ºC in temperature and 10% in relative humidity. During the test the subjects breathed through a valve (Hans Rudolph 2700, Kansas City, MO, USA) and respiratory gas exchange was determined using an automated open-circuit system (Metasys, Brainware, La Valette, France). Oxygen and CO2 content and air flow rate were recorded breath by breath. Before each trial, the system was calibrated with a mixture of O2 and CO2 of known composition (O2 15%, CO2 5%, N2 balanced) (Carburos Metálicos, Barcelona, Spain) and with ambient air. Hemodynamic information of participants was determined with non-invasive finger cuff technology (Nexfin, BMEYE Amsterdam, Netherlands). The Nexfin device provides continuous blood pressure (BP) monitoring from the resulting pulse pressure waveform, and calculates: systolic and diastolic blood pressure (SBP and DBP). Participants were connected by wrapping an inflatable cuff around the middle phalanx of the finger. The finger artery pulsing is 'fixed' to a constant volume by application of an equivalent change in pressure against the blood pressure resulting in a waveform of the pressure (clamp volume method). Electrocardiogram (ECG) was continuously monitored (DMS Systems, DMS-BTT wireless Bluetooth ECG transmitter and receiver, software DMS Version 4.0, Beijing, China). The tests were carried out at least 3 hours after a light meal and participants were instructed not to perform any vigorous physical activity for 72 hours before testing. Participants repeated this test after 6 weeks of training and after 3 weeks of detraining.

Maximal strength and power testing. Maximal strength and maximal power of upper and lower limbs, respectively, were measured (Musclelab Power System, Porsgruun, Norway) in each participant. Estimated 1 RM-chest press and 1RM-squat based on submaximal loads was calculated. In the chest press exercise the load started with 25 kg, and continued with 35 kg, 45 kg, 55 kg, 65 kg, etc. and in the squat exercise they started with 45 kg and continued with 65 kg, 85 kg, 105 kg, etc. until they could not perform 1 repetition. Based on these results the maximal 1RM was registered and the force/velocity relationship graph was plotted to determine the maximal power.

All exercise tests were carried out at least 3 hours after a light meal and participants were instructed not to perform any vigorous physical activity for 72 hours before testing. Participants repeated these tests after 6 weeks of training and after 3 weeks of detraining.

Data analysis The following maximal values of performance and cardiorespiratory variables were registered during the tests: maximal cycling workload (Wmax), maximal oxygen uptake (VO2 max), maximal expiratory ventilation per minute (VE max), maximal heart rate (HR max), maximal 1RM-squat and maximal 1RM-chest. The group means in the different conditions were compared using the non-parametric Friedman.

A PC analysis of the time series of the following selected cardiorespiratory variables: expired fraction of O2 (FeO2), expired fraction of CO2 (FeCO2), ventilation (VE), systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) was performed to obtain information about the CVCRC in each participant. The median of PC1 coefficient of congruence was obtained in each group and condition (before, after training and detraining). The null hypothesis of a constant PC congruence median over the control group and the training groups was tested through non-parametric Kruskal-Wallis. Mann Whitney U matched pairs test analysis was also performed to assess statistically significant differences between each couple of different conditions. Effect sizes (Cohen's d) were computed to demonstrate the magnitude of standardized medians' differences where effects reached p < .05 level.

ELIGIBILITY:
Inclusion Criteria:

* healthy physically active males
* physical education students
* signed an informed consent form

Exclusion Criteria:

* No confirm their healthy status
* No signed an informed consent form

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular and cardiorespiratory coupling by the principal component (PC) analysis | 3 months
  A PC analysis of the time series of the following selected cardiorespiratory variables: expired fraction of O2 (FeO2), expired fraction of CO2 (FeCO2), ventilation (VE), systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) is performed to obtain information about the CVCRC in each participant.
  (The principal component (PC) analysis is a common statistical technique that has been used to recognize such coordinative variables)
  The median of PC1 coefficient of congruence was obtained in each group and condition (before, after training and detraining) to evaluate the dimensional changes of the CVCRC before and after a period of 6 weeks of different training modalities (AT, RT and AT+RT) and 3 weeks after detraining in healthy young men.

REFERENCES:
- [Background] Friedman L, Dick TE, Jacono FJ, Loparo KA, Yeganeh A, Fishman M, Wilson CG, Strohl KP. Cardio-ventilatory coupling in young healthy resting subjects. J Appl Physiol (1985). 2012 Apr;112(8):1248-57. doi: 10.1152/japplphysiol.01424.2010. Epub 2012 Jan 19. PMID 22267392
- [Background] Garcia AJ 3rd, Koschnitzky JE, Dashevskiy T, Ramirez JM. Cardiorespiratory coupling in health and disease. Auton Neurosci. 2013 Apr;175(1-2):26-37. doi: 10.1016/j.autneu.2013.02.006. Epub 2013 Mar 13. PMID 23497744
- [Background] Wu SD, Lo PC. Cardiorespiratory phase synchronization during normal rest and inward-attention meditation. Int J Cardiol. 2010 Jun 11;141(3):325-8. doi: 10.1016/j.ijcard.2008.11.137. Epub 2009 Jan 14. PMID 19144415
- [Background] Braith RW, Stewart KJ. Resistance exercise training: its role in the prevention of cardiovascular disease. Circulation. 2006 Jun 6;113(22):2642-50. doi: 10.1161/CIRCULATIONAHA.105.584060. No abstract available. PMID 16754812
- [Background] Pollock ML, Franklin BA, Balady GJ, Chaitman BL, Fleg JL, Fletcher B, Limacher M, Pina IL, Stein RA, Williams M, Bazzarre T. AHA Science Advisory. Resistance exercise in individuals with and without cardiovascular disease: benefits, rationale, safety, and prescription: An advisory from the Committee on Exercise, Rehabilitation, and Prevention, Council on Clinical Cardiology, American Heart Association; Position paper endorsed by the American College of Sports Medicine. Circulation. 2000 Feb 22;101(7):828-33. doi: 10.1161/01.cir.101.7.828. No abstract available. PMID 10683360